CLINICAL TRIAL: NCT06906796
Title: The Effect of Diaphragmatic Breathing Exercise and Posture Exercises on Posture, Pain and Quality of Life in E-Athletes
Brief Title: The Effect of Diaphragmatic Breathing Exercise and Posture Exercises in E-Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Okan Sahin, Principal Investigator, PT, PhD (c), Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EATL-2025
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: E-Athletes
Keywords: Diaphragmatic breathing exercise; Posture exercise; Pain; Posture; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Individuals who are e-athletes between the ages of 18-30 who met the inclusion criteria will be included in the study. The study's sample size is calculated as 38 and randomized to exercise group and control groups. All evaluations of the participants will be held at Istanbul Health and Technology University Faculty of Health Sciences Manual Therapy Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Experimental): The exercise group will perform diaphragmatic breathing exercise and posture exercises 3 days a week for 6 weeks. After the diaphragmatic breathing exercise is performed for 5 minutes, individuals will perform each of the posture exercises with 10 repetitions.
  Interventions: Other: Diaphragmatic breathing exercise and posture exercises
- Control Group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Diaphragmatic breathing exercise and posture exercises — Diaphragmatic breathing exercise: Before starting the exercise protocol, individuals in the exercise group will be given training on diaphragmatic breathing exercises. During the exercise sessions, individuals will be advised to place one hand on their abdomen and the other on their chest while lying on their back and to increase abdominal movement by breathing slowly through the nose, thus decreasing rib cage movement. The diaphragmatic breathing exercise will be performed for 5 minutes.
  Posture exercises: Individuals will be given posture exercise training before starting the exercise protocol. The smoothness of the movements will be checked throughout the exercise. Chin tuck, shoulder rotation, neck extension with exercise rubber and right-left lateral flexion, pectoral stretching with hands behind, pectoral stretching in the corner and head rib cage extension exercises will be applied as posture exercises. Each exercise will be done with 10 repetitions.
  Arms: Exercise Group

SUMMARY:
There are many studies in the literature on diaphragmatic breathing exercise and posture exercises, but there are limited studies examining the effects of diaphragmatic breathing exercise and posture exercises on posture, pain and quality of life in e-athletes.

The investigators aim to contribute to the literature by examining the effects of diaphragmatic breathing exercise and posture exercises on posture, pain and quality of life in e-athletes.

DETAILED DESCRIPTION:
Electronic sports (E-sports) can be defined as a sport where individuals can play games from anywhere in the world via the internet or where people from various parts of the world play thanks to international and local organizations held at certain times. E-sports is a very popular sports field thanks to the ability to play on computer-based game systems in a globally competitive arena.

E-sports can be seen as a recreational activity outside of work hours. With its easy accessibility, area of influence and it is benefits to the individual involved, e-sports emerged as a popular recreational activity of the technology age. On the other hand, it is also considered a kind of gaming addiction. It is stated that the average gaming time is 5.2 hours per day. However, it is reported that these athletes can spend up to 14 hours per day on training or matches.

Although e-sports athletes sit at their desks for long periods during competitions, they exhibit highly coordinated movement patterns in the virtual world. The health problems seen in e-sports players are like those seen in general office workers. Musculoskeletal problems that develop due to staying in the same position for a long time can be seen in these athletes. Chronic pain that develops due to the musculoskeletal system can be shown as an example of these problems.

The increasing competitive pressure on e-sports players and the process of reaching elite performance levels can make them prone to mental health symptoms. According to research conducted on e-football players, the prevalence of mental health deterioration symptoms is high in e-football players, with 22% showing anxiety symptoms and 37% showing depression symptoms. On the other hand, e-sports players are known to have a higher prevalence of insomnia and anxiety than non-gaming participants.

Many studies have indicated that breathing exercises significantly affect both the physical and mental state of the individual. Regular practice of diaphragmatic breathing exercise leads to significant improvements in sleep quality and overall well-being, as well as reductions in respiratory rate, depression, and anxiety levels. Such exercises are deemed essential not only for the rehabilitation of patients but also for safeguarding against conditions that adversely impact the quality of life, including depression and anxiety, in healthy individuals. Scientific studies indicate that posture exercises coupled with diaphragmatic breathing exercise, positively influence pain levels and enhance quality of life.

The investigators aim to contribute to the literature by examining the effects of diaphragmatic breathing exercise and posture exercises on posture, pain and quality of life in e-athletes.

ELIGIBILITY:
Inclusion Criteria:

* Playing e-sports games for at least 1 year
* Playing a type of game played using a computer

Exclusion Criteria:

* Having any active or chronic disease
* Having a history of injury involving the musculoskeletal system
* Having a congenital/acquired mental or physical disability that would prevent participation in the study
* Having cooperation problems
* Using sleeping pills due to sleep problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
Posture Analysis | Baseline, 6th week
  Posture analysis of individuals will be done with New York Posture Rating Chart Test (NYPR). With this method, 13 different body parts are scored according to three different degrees of posture disorder. A score of 5 points is given if the person's posture is good,3 points if it is moderately impaired and 1 point if it is severely impaired, and the total score varies between 13 and 65. According to the standardized evaluation criteria developed for this assessment method, the result was indicated as 'very good' if the score was ≥45, 'good' if the score was between 40 and 44, 'fair' if the score was between 30 and 39, 'weak' if the score was between 20 and 29, and 'poor' if the score was ≤19. Higher scores indicate better postural condition. Items from this chart were used to analyse the posture of body parts for comparison between groups.
The Visual Analog Scale (VAS) | Baseline, 6th week
  This scale was used to evaluate the pain. According to the VAS, pain severity is graded as "no pain" as 0 points and "worst pain imaginable" as 10 points (10 cm scale). VAS is a reliable and valid pain measurement method in the evaluation of pain.

SECONDARY OUTCOMES:
Nottingham Health Profile | Baseline, 6th week
  The NHP is an instrument designed to measure subjective health status containing 38 items (answered ''yes'' or ''no'') that assess subjective distress in six subgroups: physical mobility (eight items), pain (eight items), sleep (five items), emotional reactions (nine items), social isolation (five items), and energy (three items). Scores for each subgroup range from 0 (no problem) to 100 (all problems listed were present).

CONTACTS AND LOCATIONS:
Overall Officials: Okan Şahin, PT, MSc, Principal Investigator — Istanbul Health and Technology University
Locations (1):
- Bahçeşehir University, Istanbul, Turkey, Turkey (Türkiye)